CLINICAL TRIAL: NCT04255199
Title: Watchful Waiting as a Strategy for Reducing Low-value Spinal Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1534721
Record Dates: First submitted 2020-01-16; First posted 2020-02-05 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Primary care and urgent care clinicians randomized to the intervention arm will receive two to three visits with a standardized patient instructor who will physicians how to facilitate patient acceptance of a watchful waiting strategy with regard to spinal imaging in the context of acute low back pain.
  Interventions: Behavioral: Intervention
- Control (Placebo Comparator): Primary care and urgent care clinicians randomized to the control arm will receive a single visit with a standardized patient who simulates a visit with patient with acute low back pain but will deliver no instruction on patient communication or other content.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Control — Clinicians randomized to the control group will receive a single visit with a standardized patient instructor (SPI) scheduled during usual office hours. SPIs will portray a patients with acute back pain but will deliver no formative training or feedback to the primary care physicians randomized to the control arm.
  Arms: Control
Behavioral: Intervention — Clinicians randomized to the intervention group will receive 2-3 visits with a standardized patient instructor (SPI) scheduled during usual office hours over ~3 month period. For intervention physicians, SPIs will portray patients with acute back pain and will provide formative feedback to physicians and specific instruction in communication techniques to facilitate patient acceptance of a watchful waiting strategy with respect to spinal imaging. The specific communication techniques and sequence will be determined based on pre-trial literature review, patient focus groups, and interviews of primary care physicians who will not participate in the trial.
  Arms: Intervention

SUMMARY:
The investigators will learn from the study whether actors playing the roles of patients (standardized patients) can help primary care and urgent care clinicians develop skill in offering watchful waiting to patients with acute low back pain as a means of averting low-value spinal imaging. Using patient and physician feedback, this study will refine and evaluate -- in a controlled experiment -- a simulated standardized patient intervention to enhance primary care physician use of watchful waiting when patients request low-value spinal imaging. The long-term goal of this study is to discover communication strategies primary care physicians can use to avert costly, potentially harmful testing while maintaining the patient-doctor relationship.

DETAILED DESCRIPTION:
Overutilization is increasingly viewed within the framework of patient safety. In primary care, patients with acute low back pain frequently request diagnostic imaging, and primary and urgent care clinicians feel pressure to acquiesce to such requests to sustain patient trust and satisfaction. Spinal imaging in patients with acute low back pain poses risks from diagnostic evaluation of false-positive findings, patient labeling and anxiety, and unnecessary treatment (including spinal surgery) with potential downstream complications.

Watchful waiting advice has been found an effective strategy to reduce low-value treatment (e.g., pediatric ear infections), and some evidence suggests a watchful waiting approach would be acceptable to many patients requesting tests. Meanwhile, psychological theory suggests that physician messages could be tailored to magnify patient acceptance of a watchful waiting strategy.

The investigators will refine and evaluate a novel simulated intervention using standardized patients (SPs) -- or actors playing the roles of patients - to teach clinicians to endorse a watchful waiting approach when patients request low-value spinal imaging for low back pain. Specific aims are:

Aim 1: To use key informant interviews of front-line clinicians and focus groups with primary care patients to refine a theory-informed standardized patient-based intervention designed to teach practicing clinicians how to advise watchful waiting when patients request low-value spinal imaging for low back pain.

Aim 2: To test the effectiveness of standardized patient instructor (SPI)-delivered clinician training in the use of watchful waiting in a randomized clinical trial.

The investigators hypothesize that the intervention will: a) reduce rates of low-value spinal imaging among actual patients with acute back pain seen by clinicians post-intervention (adjusting for pre-trial rates); b) increase clinician advice to pursue watchful waiting during a followup visit with an unannounced SP; c) increase clinician self-reported use and efficacy of advising watchful waiting with actual low back pain patients; and d) have no adverse impact on actual patient trust and satisfaction with physicians; and e) reduce rates of neck imaging (among neck pain patients) and overall diagnostic testing (among all adult patients).

Aim 3: To assess whether the intervention effects generalize to other low-value imaging tests and diagnostic tests in general.

The investigators hypothesize that the SP intervention will: a) decrease rates of neck imaging among actual patients with neck pain seen by study clinicians during the follow-up period (adjusting for baseline rates); b) decrease rates of overall diagnostic tests among all adult patient seen by study clinicians during the follow-up period (adjusting for baseline rates); and c) increase PCP self-reported use and efficacy of advising watchful waiting for patients with neck pain, other musculoskeletal pain, and other non-musculoskeletal somatic complaints.

ELIGIBILITY:
Inclusion Criteria: Primary care and urgent care clinicians in the two health systems will be eligible if:

1. they intend to practice either at least 50% full-time equivalent (FTE) adult primary or urgent care in one of the target clinics for the trial duration
2. they have been in active full-time or 50% FTE practice within the health system for at least two years prior to enrollment (to enable collection of baseline testing rates).
3. Nurse practitioners and physicians assistants will be eligible if they practice in the capacity of a primary care or urgent care clinicians and meet the other requirement above.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Adjusted rate of spinal imaging during 18-month follow-up | 18 months following date of first SPI visit
  Rate of lumbar spinal x-ray, CT, or MRI during follow-up period, adjusted for imaging rate during 12 month pre-randomization period

SECONDARY OUTCOMES:
Adjusted rate of advanced spinal imaging during 18-month follow-up | 18 months following date of first SPI visit
  Rate of lumbar CT or MRI during follow-up period, adjusted for imaging rate during 12 month pre-randomization period
Adjusted rate of lumbar x-ray imaging during 18-month follow-up | 18 months following date of first SPI visit
  Rate of lumbar x-ray during follow-up period, adjusted for imaging rate during 12 month pre-randomization period
Use of watchful waiting communication techniques based on coded transcripts | 6 months post-intervention
  Using transcripts of audio-recordings of a single post-intervention SP visit per randomized physician, investigators will identify physicians' use of communication techniques targeted by the intervention based on coding conducted by trained research assistants. Communication techniques will be identified based on a coding manual that will be developed by the investigators using transcripts of baseline standardized patient visits prior to instruction. The outcome will be a count of targeted communication techniques used during the follow-up visits. Investigators will report the relative rate of technique use adjusted for counts of techniques used during baseline standardized patient visits.
Physician self-reported use of watchful waiting techniques in post-intervention questionnaires | 6 months post-intervention
  Study physicians will complete an on-line survey 6 months after final SPI visits and will report the frequency of use of watchful waiting techniques on Likert scales created by the investigators for this project.
Adjusted rate of neck imaging during 18-month follow-up | 18 months following date of first SPI visit
  Rate of neck x-ray, CT, or MRI during follow-up period, adjusted for imaging rate during 12 month pre-randomization period
Adjusted rate of diagnostic test ordering during 18-month follow-up | 18 months following date of first SPI visit
  Rate of diagnostic test ordering (laboratory, imaging, cardiac, gastrointestinal and vascular tests) during 18 month follow-up period, adjusted for diagnostic test ordering rate during 12 month pre-randomization period
Patient experience ratings during 18-month follow-up | 18 months following date of first SPI visit
  Mean difference (vs. baseline period) in percent of patients rating clinicians either 9 or 10 on the Consumer Assessment of Healthcare Providers and Systems Overall Doctor Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Joshua J Fenton, MD, MPH, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Center for Healthcare Policy and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data would be shared with other researchers if their research protocols were institutional review board approved, and our team had sufficient time and resources to generate the individual participant data for secure data transfer.

REFERENCES:
- [Background] Fenton JJ, Jerant A, Franks P, Gosdin M, Fridman I, Cipri C, Weinberg G, Hudnut A, Tancredi DJ. Watchful waiting as a strategy to reduce low-value spinal imaging: study protocol for a randomized trial. Trials. 2021 Feb 27;22(1):167. doi: 10.1186/s13063-021-05106-x. PMID 33639993
- [Result] Fenton JJ, Cipri C, Gosdin M, Tancredi DJ, Jerant A, Robinson CA, Xing G, Fridman I, Weinberg G, Hudnut A. Standardized Patient Communication and Low-Value Spinal Imaging: A Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2441826. doi: 10.1001/jamanetworkopen.2024.41826. PMID 39504026